CLINICAL TRIAL: NCT05496309
Title: Causes and Mechanisms of Space Hemolysis At High Altitudes (ANEMIA)
Brief Title: Causes and Mechanisms of Space Hemolysis At High Altitudes
Acronym: ANEMIA
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Guy Trudel, Professor of Medicine, Surgery and Biochemistry, Ottawa Hospital Research Institute
Other Study IDs: 0220470-01H
Record Dates: First submitted 2022-07-28; First posted 2022-08-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Anemia; Weightlessness
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: The group is a cohort of 4 persons.

SUMMARY:
Anemia is a lack of red blood cells (RBCs) in the circulation. Because RBCs carry the oxygen your body needs to function, anemia can affect one's ability to stay awake, alert, and perform physical activities. Anemia may happen for several reasons, including increased RBC destruction. Anemia often occurs in people who have been in bed for long periods (e.g., if they are very sick) or have decreased mobility (anemia of immobility). Interestingly, astronauts who have left Earth and traveled in space also return anemic. In fact, 5 decades of NASA data showed that astronauts' anemia was more severe the longer they were in space. In another study, astronauts aboard the International Space Station were shown to destroy 54% more of their RBCs in space. RBC destruction may be the culprit of space anemia as well as anemia of immobility on Earth. The ANEMIA Study proposes to measure key aspects of RBC destruction in astronauts in space. These measures will test critical hypotheses on the effects of spaceflight on red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Astronauts selected to fly on a space mission.

Exclusion Criteria:

* Astronauts not selected to fly on a space mission.

Ages: 24 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Astronauts selected to fly on a space mission.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Hemolysis in astronauts is assessed using exhaled breath samples. | Before spaceflight.
Change from baseline hemolysis in astronauts is assessed during spaceflight using exhaled breath samples. | Baseline and during spaceflight.
Change from baseline hemolysis in astronauts is assessed after spaceflight, up to 1 month, using exhaled breath samples. | After spaceflight, up to 1 month.
Hemolysis in astronauts is assessed using blood markers CBC, reticulocytes, haptoglobin, bilirubin (total+direct), LDH, ferritin, iron, and TIBC. | Before spaceflight.
Change from baseline hemolysis in astronauts is assessed during spaceflight using blood markers CBC, reticulocytes, haptoglobin, bilirubin (total+direct), LDH, ferritin, iron, and TIBC. | Baseline and during spaceflight.
Change from baseline hemolysis in astronauts is assessed after spaceflight, up to 1 month, using blood markers CBC, reticulocytes, haptoglobin, bilirubin (total+direct), LDH, ferritin, iron, and TIBC. | After spaceflight, up to 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Trudel, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
There may be multiauthor publication involving multiple PI on the same astronauts for this mission. Each PI contributing to the manuscript their individual data.